CLINICAL TRIAL: NCT03531437
Title: Comparison of Coagulation Profiles in Oral Contraceptive Pills Users Between 1.5 mg Estradiol/2.5 mg Nomegestrol Acetate (Zoely) and 15 mcg Ethinylestradiol/60 mcg Gestodene (Minidoz): A Randomized Control Trial
Brief Title: Comparison of Coagulation Profiles Between Zoely and Minidoz: RCT
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: problem with recruiting participants
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Nalinee Panichyawat, Siriraj hospital, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 656/2558 (Si726/2015)
Record Dates: First submitted 2016-01-11; First posted 2018-05-21 (Actual); Last update posted 2018-05-21 (Actual); Status verified 2018-05

CONDITIONS: Contraception; Hypercoagulability
MeSH Terms: conditions — Thrombophilia | interventions — Estradiol; nomegestrol acetate; Ethinyl Estradiol; Gestodene

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Zoely (Active Comparator): Monophasic combined oral contraceptive pills 24 white active tablets and 4 yellow inactive tablets each active tablet contains 1.5 mg estradiol and 2.5 mg nomegestrol acetate 3 cycles
  Interventions: Drug: 1.5 mg estradiol and 2.5 mg nomegestrol acetate
- Minidoz (Active Comparator): Monophasic combined oral contraceptive pills 24 active tablets and 4 inactive tablets each active tablet contains ethinylestradiol 15 µg and gestodene 60 µg 3 cycles
  Interventions: Drug: 15 µg ethinylestradiol and 60 µg gestodene

INTERVENTIONS:
Drug: 1.5 mg estradiol and 2.5 mg nomegestrol acetate
  Other Names: Zoely®
  Arms: Zoely
Drug: 15 µg ethinylestradiol and 60 µg gestodene
  Other Names: Minidoz®
  Arms: Minidoz

SUMMARY:
The purpose of this study is to compare the effects of Zoely® and Minidoz® on hemostatic profiles

DETAILED DESCRIPTION:
compare the effects of Zoely® and Minidoz® on hemostatic profiles : D-dimer, Antithrombin and fibrinogen

ELIGIBILITY:
Inclusion Criteria:

* Woman age 19-40 yr
* Normal uterus and both adnexae
* BMI < 28.5 kg/m2
* Require contraception with COCs

Exclusion Criteria:

* Pregnancy
* Postartum period within 6 wk
* Smoking
* BP ≥ 140/90 mmHg
* Contraindication to COCs : VTE, cerebrovascular disease, cardiovascular disease, migraine with aura, hepatitis, undiagnosed abnormal uterine bleeding, CA breast, DM with DN/DR
* use of liver-enzyme-inducing drugs, drugs affecting the haemostatic system
* Use contraceptive steroids within 3 months

Ages: 19 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 112 (Actual)
Dates: Start 2016-03; Primary Completion 2018-01 (Actual); Study Completion 2018-04-18 (Actual)

PRIMARY OUTCOMES:
D-dimer | 12 weeks
  µg/L

SECONDARY OUTCOMES:
fibrinogen | 12 weeks
  mg/dL
antithrombin III | 12 weeks
  percent
to access menstrual cycle and bleeding pattern, side effects of Zoely® and Minidoz® | 12 weeks

IPD SHARING:
Plan to Share IPD: Undecided